CLINICAL TRIAL: NCT00253448
Title: Phase II Trial of Conventional Radiotherapy With Stereotactic Radiosurgery to High Risk Tumor Regions as Determined by Functional Imaging in Patients With Glioblastoma Multiforme
Brief Title: Stereotactic Radiosurgery and Radiation Therapy in Treating Patients With Glioblastoma Multiforme
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CWRU1302; P30CA043703 (NIH); CASE-CWRU-1302 (Other: Case Comprehensive Cancer Center)
Record Dates: First submitted 2005-11-11; First posted 2005-11-15 (Estimated); Results first posted 2011-07-26 (Estimated); Last update posted 2011-08-29 (Estimated); Status verified 2011-08

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: adult glioblastoma; adult giant cell glioblastoma; adult gliosarcoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Glioblastoma; Gliosarcoma | interventions — Radiotherapy; Radiosurgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Radiation: radiation therapy — No more than 2 weeks later, patients undergo conventional radiotherapy once daily, 5 days a week, for 6 weeks.
Radiation: stereotactic radiosurgery — stereotactic radiosurgery to high-risk areas of active tumor determined by MR-spectroscopy

SUMMARY:
RATIONALE: Stereotactic radiosurgery may be able to send x-rays directly to the tumor and cause less damage to normal tissue. Radiation therapy uses high-energy x-rays to kill tumor cells. Giving stereotactic radiosurgery together with radiation therapy may kill more tumor cells.

PURPOSE: This phase II trial is studying how well giving stereotactic radiosurgery together with radiation therapy works in treating patients with glioblastoma multiforme.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the feasibility and efficacy of stereotactic radiosurgery to high-risk tumor regions and conventional radiotherapy in patients with glioblastoma multiforme.
* Determine overall survival of patients treated with this regimen.

Secondary

* Determine 6-month progression-free survival of patients treated with this regimen.
* Determine the absence of tumor growth and/or activity on conventional MR/MR spectroscopy imaging in patients treated with this regimen.
* Determine the frequency and severity of RTOG (Radiation Therapy Oncology Group) CNS toxic effects in patients treated with this regimen.
* Determine the neurologic function and quality of life of patients treated with this regimen.

OUTLINE: This is a pilot study.

Patients undergo stereotactic radiosurgery to high-risk areas of active tumor determined by MR-spectroscopy. No more than 2 weeks later, patients undergo conventional radiotherapy once daily, 5 days a week, for 6 weeks.

Quality of life is assessed at baseline, weekly during radiotherapy, at 1 and 3 months after completion of radiotherapy, and then every 3 months for 2 years, every 6 months for 3 years, and annually thereafter.

After completion of study treatment, patients are followed periodically for at least 5 years.

PROJECTED ACCRUAL: A total of 35 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed grade IV malignant glioblastoma multiforme

  * Diagnosis by surgical biopsy or resection within the past 5 weeks
* Post-operative diagnostic contrast-enhanced MRI scan with MR spectroscopy must be performed prior to initiating study treatment

  * High-risk area of active tumor without margin by MR spectroscopy

    * Meets the following criteria for radiosurgery:

      * Maximum diameter ≤ 40 mm
      * Located > 5 mm from the optic nerve or chiasm
      * Does not involve the brainstem
* No multifocal or recurrent malignant glioma

PATIENT CHARACTERISTICS:

Performance status

* Karnofsky 50-100%

Life expectancy

* At least 3 months

Hematopoietic

* Not specified

Hepatic

* Not specified

Renal

* Not specified

Other

* Not pregnant
* Negative pregnancy test

PRIOR CONCURRENT THERAPY:

Chemotherapy

* At least 6 weeks since chemotherapy
* Concurrent chemotherapy allowed

Endocrine therapy

* Concurrent steroids allowed, but at the smallest therapeutic dose possible

Radiotherapy

* No prior in-field radiotherapy to the head and neck

Surgery

* See Disease Characteristics
* Recovered from prior surgery or any post-operative complication

Other

* Concurrent antiseizure medications allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2002-12; Primary Completion 2009-12 (Actual); Study Completion 2011-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Einstein, MD, PhD, Principal Investigator — Kettering Medical Center, Wright State University
Locations (2):
- United States (2):
  - Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio
  - Southwest General Health Center, Cleveland, Ohio

REFERENCES:
- [Derived] Einstein DB, Wessels B, Bangert B, Fu P, Nelson AD, Cohen M, Sagar S, Lewin J, Sloan A, Zheng Y, Williams J, Colussi V, Vinkler R, Maciunas R. Phase II trial of radiosurgery to magnetic resonance spectroscopy-defined high-risk tumor volumes in patients with glioblastoma multiforme. Int J Radiat Oncol Biol Phys. 2012 Nov 1;84(3):668-74. doi: 10.1016/j.ijrobp.2012.01.020. Epub 2012 Mar 22. PMID 22445005

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects recruited from 12/31/2002 to 5/8/2008 from medical clinic
Pre-assignment Details: One patient was not eligible for unknown reason
Groups:
- Stereotactic Radiosurgery Plus Conventional Radiotherapy: Single 15-24 Gy Gamma Knife radiosurgical treatment to MR-Spectroscopy active region followed by 60 Gy of conventionally fractionated radiotherapy (2.0 Gy will be given daily 5 days per week for a total of 60.0 Gy)
Period: Overall Study
Arm/Group | Stereotactic Radiosurgery Plus Conventional Radiotherapy
Started | 35
Completed | 34
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Stereotactic Radiosurgery Plus Conventional Radiotherapy
Number analyzed (Participants) | 35
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 20
  >=65 years | 15
Age Continuous [Mean (Standard Deviation); unit: years] | 60.9 (12.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 35

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival After Treatment
Description: Followed every 3 months for 2 years, every 6 months for 3 years, and annually thereafter for at least 5 years
Time Frame: Minimum of 5 years.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Stereotactic Radiosurgery Plus Conventional Radiotherapy
Number analyzed (Participants) | 35
months
  Entire Cohort | 15.8 [11 to 19.9]
  RTOG Glioma Recursive Partitioning Class 3 n=4 | 22 [22 to 22]
  RTOG Glioma Recursive Partitioning Class 4 n=13 | 18.7 [14.5 to 29.1]
  RTOG Glioma Recursive Partitioning Class 5 n=16 | 12.5 [9.2 to 18.5]
  RTOG Glioma Recursive Partitioning Class 6 n=2 | 3.9 [2.7 to 5.1]
  Patients receiving concurrent chemotherapy | 20.8 [14.2 to 29.1]
  Patients who were not candidates for chemotherapy | 11 [7.2 to 18.5]

ADVERSE EVENTS:
Arm/Group | Stereotactic Radiosurgery Plus Conventional Radiotherapy
Serious Adverse Events (participants affected / at risk) | 4/35
Other Adverse Events (participants affected / at risk) | 0/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stereotactic Radiosurgery Plus Conventional Radiotherapy (N=35)
CVA (Nervous system disorders) | 1 (1) — Cerebrovascular Accident in a patient taking anticoagulant warfarin
Re-operation for radiation necrosis (Nervous system disorders) | 3 (3) — Re-operation for neurological symptom progression secondary to radiation necrosis

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes